CLINICAL TRIAL: NCT01830556
Title: Cetuximab 5-FU and Cisplatin or Carboplatin Versus Cetuximab With Paclitaxel and Carboplatin Treatment of Metastatic Squamous Cell Carcinoma of Head and Neck
Brief Title: Randomised Phase II, Cetuximab in Combination With 5FU and Cisplatin or Carboplatin Versus Cetuximab in Combination With Paclitaxel and Carboplatin for Treatment of Patients With Metastatic Squamous Cell Carcinoma of the Head and Neck
Acronym: CETMET
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Karolinska University Hospital (Other)
Responsible Party: Principal Investigator, Signe Friesland, MD, PhD, Karolinska University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CETMET study
Record Dates: First submitted 2013-04-10; First posted 2013-04-12 (Estimated); Last update posted 2013-05-21 (Estimated); Status verified 2013-05

CONDITIONS: Squamous Cell Carcinoma of the Head and Neck
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck | interventions — Cetuximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm A: cetuximab with 5FU and carboplatin or cisplatin (Active Comparator): Arm A:Day 1 Cetuximab 400 mg/m2 iv 120 minutes Day 8 and 15 Cetuximab 250 mg/m2 iv 60 minutes Day 1 Cisplatin 100mg/m2 or Carboplatin AUC 5 day 1-4 5-Fluorouracil 1000 mg/m2 iv 24 h maintenance treatment thereafter with cetuximab 500 mg/m2 every second week until PD or toxicity
  Interventions: Drug: Cetuximab
- Arm B: cetuximab paclitaxel and carboplatin (Experimental): Arm B day 1 Cetuximab 400 mg/m2 iv 120 minutes Day 8 and 15 Cetuximab 250 mg/m2 iv 60 minutes day 1 Paclitaxel 175 mg/m2 day 1 Carboplatin AUC 5 treatment for 6 cycles thereafter maintenance treatment day 1 Cetuximab 500 mg/m2 every second week treatment until progress or unacceptable toxicity
  Interventions: Drug: Cetuximab

INTERVENTIONS:
Drug: Cetuximab — Group A:Day 1 Cetuximab 400 mg/m2 iv 120 minutes Day 8 and 15 Cetuximab 250 mg/m2 iv 60 minutes Day 1 Cisplatin 100mg/m2 or Carboplatin AUC 5 day 1-4 5-Fluorouracil 1000 mg/m2 iv 24 h Group B day 1 Cetuximab 400 mg/m2 iv 120 minutes Day 8 and 15 Cetuximab 250 mg/m2 iv 60 minutes day 1 Paclitaxel 175 mg/m2 day 1 Carboplatin AUC 5 treatment for 6 cycles thereafter day 1 Cetuximab 500 mg/m2 every second week treatment until progress or unacceptable toxicity
  Other Names: Erbitux

SUMMARY:
Primary To investigate in patients with relapsed or metastatic squamous cell carcinoma of the head and neck whether progression free survival (PFS) in the arm with cetuximab, paclitaxel and carboplatin based chemotherapy is not markedly worse than PFS in the arm with cetuximab and 5-FU, cisplatin or carboplatin based chemotherapy.

Secondary

To compare in patients with relapsed or metastatic squamous cell carcinoma of the head and neck the following study variables between both treatment arms:

* Best overall response
* Duration of response
* Time to treatment failure
* Overall survival
* Safety

DETAILED DESCRIPTION:
Recurrent and/or metastatic SCCHN patients are, by definition patients with recurrent disease and/or with newly diagnosed distant metastases, although this group of patients has a very heterogeneous disease characteristic, they share a dismal prognosis that has changed little in the past 30 years. The median survival time remains around 6-8 months with a poor quality of life. Patients with resectable locoregionally recurrent SCCHN may benefit from surgery. Patients with recurrent SCCHN who are not suitable for curative salvage surgery or re-irradiation, and patients who have distant metastases, usually receive CT (Cohen EE et al.) A number of compounds demonstrate single-agent activity in recurrent and/or metastatic disease including cisplatin, carboplatin, methotrexate, 5-FU, bleomycin and the taxanes ( Scantz SP et al). Cisplatin is one of the most active agents identified for head and neck cancer, with carboplatin providing an alternative for patients unable to tolerate cisplatin. While carboplatin is associated with lower response rates than cisplatin, there appears to be no difference between the agents in terms of survival

Cetuximab is a targeted therapeutic agent, a chimeric IgG1 monoclonal antibody that specifically binds to the EGFR with high affinity, internalising the receptor and preventing the ligands EGF and TGF-alfa from interacting with the receptors and thus effectively blocking ligand-induced EGFR phosphorylation. In addition, cetuximab has been found to potentiate the effects of chemotherapy and radiotherapy in experimental systems. The dose of cetuximab has been found to be generally safe and effective in several studies in major tumor types expressing the EGFR. These included colorectal cancer, squamous cell carcinoma of the head and neck and non-small cell lung cancer, with cetuximab given either in combination studies with chemotherapy and radiotherapy or as monotherapy. The main side effects of cetuximab monotherapy are hypersensitivity- and acne-like skin reactions.

ELIGIBILITY:
Inclusion criteria

* >18 years
* Histologically or cytologically confirmed SCCHN, relapsed and/or metastatic
* Patient must have a life expectancy of at least 3 months allowing adequate follow-up toxicity evaluation.
* Clinical examination
* 1 unidimensional lesion according to RECIST 1.1.
* PS WHO 0-1 at study entry
* Adequate hematological function defined as WBC ≥3 x 109/litre and platelets ≥100 x 109/litre, ANC > 1.5 x 109/litre and Hb > 100 g/L
* Adequate liver function; bilirubin < 1.5 x UNL, ALAT or ASAT<3.0 UNL, alkaline phosphates < 2.5 UNL.
* Creatinine clearance > 50mL/min
* Written informed consent must be obtained according to the local Ethics committee.

Exclusion Criteria:

* > 75 years
* Nasopharyngeal cancer and cancer of the paranasal sinuses
* Inability to follow the treatment and evaluation schedule
* Any other condition or therapy which in the investigator's opinion may pose a risk to the patient or interfere with the study objectives
* Pregnant or nursing females or male or female of child-bearing potential not using adequate methods of birth-control
* Patients with active infections or any other serious underlying medical condition, which would impair the ability of the patients to receive the protocol treatment
* Known hypersensitivity to any of the components of the treatment
* Legal incapacity
* Clinically significant cardiovascular disease, e.g. cardiac failure of New York Heart Association classes III-IV, uncontrolled coronary artery disease, cardiomyopathy, uncontrolled arrhythmia, uncontrolled hypertension, or history of myocardial infarction in the last 12 months.
* Patients with clinically relevant neuropathy
* Previously treated for relapsed or metastatic SCCHN except radiotherapy for previously treated relapse if terminated > 3 months before start of treatment.
* Previously treated with cetuximab, cisplatin/carboplatin, 5-FU or taxanes for locally advanced SCCHN within 3 months before study entry.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2011-11; Primary Completion 2013-11 (Estimated); Study Completion 2015-11 (Estimated)

PRIMARY OUTCOMES:
Progression free survival | 3 years
  To investigate in patients with relapsed or metastatic squamous cell carcinoma of the head and neck whether progression free survival (PFS) in the arm with cetuximab, paclitaxel and carboplatin based chemotherapy is not markedly worse than PFS in the arm with cetuximab and 5-FU, cisplatin or carboplatin based chemotherapy.

SECONDARY OUTCOMES:
Best overall response | 3 years
  To compare in patients with relapsed or metastatic squamous cell carcinoma of the head and neck the following study variables between both treatment arms:
  * Best overall response
  * Duration of response
  * Time to treatment failure
  * Overall survival
  * Safety

CONTACTS AND LOCATIONS:
Overall Officials: Signe Friesland, MD Phd, Principal Investigator — Karolinska Universityhospital
Locations (5):
- Lena Specht, Copenhagen, Denmark
- Sweden (4):
  - Karolinska Universityhospital, Stockholm, Stockholm County
  - Hedda Haugen, Gothenburg
  - Karin Söderström, Umeå
  - Akademiska Universityhospital, Uppsala